CLINICAL TRIAL: NCT07389993
Title: Diaphragm Characteristics and Respiratory Muscle Function in Parous Women With and Without Diastasis Recti Abdominis
Brief Title: Diaphragm and Breathing Muscle Characteristics in Women With and Without Diastasis Recti Abdominis After Childbirth
Acronym: DRA-DIAPH
Status: Recruiting | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Anastasia Skoura, Principal Investigator, University of Patras
Other Study IDs: DRA-DIAPHRAGM-PILOT
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diastasis Recti Abdominis (DRA)
Keywords: diastasis recti; diaphragm; RUSI; inspiratory muscle strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with diastasis recti abdominis: Parous women diagnosed with diastasis recti abdominis using a standardised ultrasonographic assessment to measure the inter-recti distance (IRD).
  Interventions: Diagnostic Test: Ultrasonographic assessment of the diaphragm; Diagnostic Test: Inspiratory muscle testing
- Women without diastasis recti abdominis: Parous women without diastasis recti abdominis, as confirmed by standardized ultrasonographic assessment of inter-recti distance (IRD).
  Interventions: Diagnostic Test: Ultrasonographic assessment of the diaphragm; Diagnostic Test: Inspiratory muscle testing

INTERVENTIONS:
Diagnostic Test: Ultrasonographic assessment of the diaphragm — Rehabilitative ultrasound imaging (RUSI) to assess diaphragm thickness and excursion under specific respiratory maneuvers.
Diagnostic Test: Inspiratory muscle testing — A standardized inspiratory muscle strength testing procedure using a POWERbreathe KH2 device to assess maximal inspiratory pressure (MIP), S-Index and peak inspiratory flow (PIF).

SUMMARY:
Diastasis Recti Abdominis (DRA) is a common condition experienced postpartum, in which the abdominal muscles separate along the midline of the abdomen due to stretching and thinning of the linea alba. It's a common condition, affecting 66-100% of women post-birth and may be associated with changes in abdominal support, posture, breathing, and trunk function. Although DRA primarily affects the muscles of the abdominal wall, it is speculated that other muscles controlling and stabilizing the trunk, such as the pelvic floor muscles or the diaphragm, might be affected as well. Currently, several studies have investigated the possible negative effects of DRA on pelvic floor function. However, little is known about how it may be related to diaphragm function and accessory breathing muscles.

The purpose of this observational study is to compare diaphragm characteristics and function, and accessory breathing muscle strength in women who have given birth, with and without DRA.

To make this possible, adult parous women from the broader Achaia region are assessed and allocated into two predefined groups based on the presence or absence of DRA. Participants undergo a single assessment session including rehabilitative ultrasound imaging (RUSI) of the diaphragm and standardized tests of inspiratory muscle strength. Additional demographic and clinical information related to pregnancy and physical activity is also recorded. The main hypothesis of this study is that women with DRA demonstrate altered diaphragm function, as well as reduced inspiratory muscle strength, compared to women without DRA. The study aims to improve understanding of the possible relationship between DRA and breathing function after childbirth and to support future research and rehabilitation approaches for women with the condition.

DETAILED DESCRIPTION:
Diastasis recti abdominis (DRA) is a common postpartum condition, characterized by stretching and thinning of the linea alba and separation of the two rectus abdominis muscles along the midline of the abdomen. Beyond cosmetic concerns, DRA has been associated with impaired abdominal wall function, altered trunk stability, and potential changes in respiratory mechanics due to the close anatomical and functional relationship between the abdominal muscles and the diaphragm.

The diaphragm plays a central role in respiration and trunk stabilization, working synergistically with the abdominal wall to regulate intra-abdominal pressure (IAP) and postural control. Alterations in abdominal wall integrity, such as those observed in DRA, may therefore influence diaphragm function and mobility, as well as overall respiratory muscle performance. However, evidence regarding the relationship between DRA and diaphragm function currently remains limited.

This observational, cross-sectional study aims to examine diaphragm characteristics and inspiratory muscle strength in parous women with and without DRA. Participants are allocated into two predefined groups according to the presence or absence of DRA, based on a standardized imaging assessment.

Diaphragm function is assessed using rehabilitative ultrasound imaging (RUSI) techniques, performed by a trained physiotherapist, following standardized procedures. Ultrasound images are obtained during specific breathing maneuvers to determine diaphragm thickness and excursion. Inspiratory muscle strength is assessed using a standardized procedure to test maximal inspiratory pressure (MIP), S-Index and Peak Inspiratory Pressure (PIF) using a POWERbreathe KH2 device. All measurements are conducted during a single assessment session, and are led by three experienced physiotherapists. Furthermore, demographic data and relevant obstetric and clinical characteristics, such as age, body mass index (BMI), parity, and time since last delivery, are recorded to describe the study population.

The study aims to explore whether women with DRA demonstrate differences in diaphragm-related parameters and inspiratory muscle strength compared with women without DRA. By improving understanding of the interaction between the abdominal wall and respiratory muscles after childbirth, this research may contribute to the development of more targeted assessment strategies and rehabilitation approaches in postpartum care.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Aged 18 to 50 years
* Parous women (at least one previous childbirth)
* At least 6 months postpartum at the time of assessment (and within 5 years postpartum)
* Ability to understand and communicate in Greek
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Current pregnancy
* Delivery within the previous 6 months
* History of severe chronic respiratory disease (e.g., chronic obstructive pulmonary disease, chronic bronchitis, pulmonary emphysema, pulmonary fibrosis)
* Presence of connective tissue disorders
* Presence of neurological disorders
* Severe musculoskeletal conditions that could affect trunk or respiratory function or limit participation in testing procedures (severe low back pain, sciatica etc.)
* Previous abdominal surgery, with the exception of cesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Parous adult women from the local community (broader Achaia region) recruited through invitations and referrals and assessed in a clinical research setting.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Inspiratory diaphragm thickness | Baseline
  Diaphragm thickness measured via ultrasound in cm at the end of a full inspiration at a standardized anatomical location.
Expiratory diaphragm thickness | Baseline
  Diaphragm thickness measured via ultrasound in cm at the end of a full expiration at a standardized anatomical location.
Diaphragm excursion | Baseline
  Diaphragm excursion measured via ultrasound in cm during quiet respiration at 60% of inspiratory capacity (IC).

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | Baseline
  Maximal Inspiratory Pressure (MIP) measured during a forceful inspiratory effort in cmΗ2Ο, using the POWERbreathe KH2 device.
S-Index | Baseline
  S-Index, a strength estimate measured in cmH2O during a forceful inspiration performed using the POWERbreathe KH2 device.
Peak Inspiratory Flow (PIF) | Baseline
  Peak Inspiratory Flow (PIF) measured in L/sec, during the same forceful inspiratory maneuver as SIndex, using the POWERbreathe KH2 device.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, PhD, Principal Investigator — University of Patras
Locations (1):
- Laboratory of Clinical Rehabilitation and Research (CPRlab), University of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beer GM, Schuster A, Seifert B, Manestar M, Mihic-Probst D, Weber SA. The normal width of the linea alba in nulliparous women. Clin Anat. 2009 Sep;22(6):706-11. doi: 10.1002/ca.20836. PMID 19637295
- [Background] Benjamin DR, Frawley HC, Shields N, van de Water ATM, Taylor NF. Relationship between diastasis of the rectus abdominis muscle (DRAM) and musculoskeletal dysfunctions, pain and quality of life: a systematic review. Physiotherapy. 2019 Mar;105(1):24-34. doi: 10.1016/j.physio.2018.07.002. Epub 2018 Jul 24. PMID 30217494
- [Background] Skoura A, Billis E, Papanikolaou DT, Xergia S, Tsarbou C, Tsekoura M, Kortianou E, Maroulis I. Diastasis Recti Abdominis Rehabilitation in the Postpartum Period: A Scoping Review of Current Clinical Practice. Int Urogynecol J. 2024 Mar;35(3):491-520. doi: 10.1007/s00192-024-05727-1. Epub 2024 Feb 10. PMID 38340172
- [Background] Mota P, Pascoal AG, Carita AI, Bo K. Normal width of the inter-recti distance in pregnant and postpartum primiparous women. Musculoskelet Sci Pract. 2018 Jun;35:34-37. doi: 10.1016/j.msksp.2018.02.004. Epub 2018 Feb 20. PMID 29494833
- [Background] Hills NF, Graham RB, McLean L. Comparison of Trunk Muscle Function Between Women With and Without Diastasis Recti Abdominis at 1 Year Postpartum. Phys Ther. 2018 Oct 1;98(10):891-901. doi: 10.1093/ptj/pzy083. PMID 30011041
- [Background] Gluppe S, Ellstrom Engh M, Kari B. Women with diastasis recti abdominis might have weaker abdominal muscles and more abdominal pain, but no higher prevalence of pelvic floor disorders, low back and pelvic girdle pain than women without diastasis recti abdominis. Physiotherapy. 2021 Jun;111:57-65. doi: 10.1016/j.physio.2021.01.008. Epub 2021 Feb 13. PMID 33691943
- [Background] Boussuges A, Rives S, Finance J, Bregeon F. Assessment of diaphragmatic function by ultrasonography: Current approach and perspectives. World J Clin Cases. 2020 Jun 26;8(12):2408-2424. doi: 10.12998/wjcc.v8.i12.2408. PMID 32607319
- [Background] Kolar P, Sulc J, Kyncl M, Sanda J, Cakrt O, Andel R, Kumagai K, Kobesova A. Postural function of the diaphragm in persons with and without chronic low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):352-62. doi: 10.2519/jospt.2012.3830. Epub 2011 Dec 21. PMID 22236541
- [Background] Hodges P, Kaigle Holm A, Holm S, Ekstrom L, Cresswell A, Hansson T, Thorstensson A. Intervertebral stiffness of the spine is increased by evoked contraction of transversus abdominis and the diaphragm: in vivo porcine studies. Spine (Phila Pa 1976). 2003 Dec 1;28(23):2594-601. doi: 10.1097/01.BRS.0000096676.14323.25. PMID 14652476
- [Background] Hodges PW, Butler JE, McKenzie DK, Gandevia SC. Contraction of the human diaphragm during rapid postural adjustments. J Physiol. 1997 Dec 1;505 ( Pt 2)(Pt 2):539-48. doi: 10.1111/j.1469-7793.1997.539bb.x. PMID 9423192
- [Background] Hodges PW, Cresswell AG, Daggfeldt K, Thorstensson A. In vivo measurement of the effect of intra-abdominal pressure on the human spine. J Biomech. 2001 Mar;34(3):347-53. doi: 10.1016/s0021-9290(00)00206-2. PMID 11182126
- [Background] Hodges PW, Eriksson AE, Shirley D, Gandevia SC. Intra-abdominal pressure increases stiffness of the lumbar spine. J Biomech. 2005 Sep;38(9):1873-80. doi: 10.1016/j.jbiomech.2004.08.016. PMID 16023475
- [Background] Hodges PW, Gandevia SC. Changes in intra-abdominal pressure during postural and respiratory activation of the human diaphragm. J Appl Physiol (1985). 2000 Sep;89(3):967-76. doi: 10.1152/jappl.2000.89.3.967. PMID 10956340
- [Background] Hodges PW, Gandevia SC, Richardson CA. Contractions of specific abdominal muscles in postural tasks are affected by respiratory maneuvers. J Appl Physiol (1985). 1997 Sep;83(3):753-60. doi: 10.1152/jappl.1997.83.3.753. PMID 9292460
- [Background] Hodges PW, Heijnen I, Gandevia SC. Postural activity of the diaphragm is reduced in humans when respiratory demand increases. J Physiol. 2001 Dec 15;537(Pt 3):999-1008. doi: 10.1111/j.1469-7793.2001.00999.x. PMID 11744772
- [Background] Hodges PW, Sapsford R, Pengel LH. Postural and respiratory functions of the pelvic floor muscles. Neurourol Urodyn. 2007;26(3):362-71. doi: 10.1002/nau.20232. PMID 17304528
- [Background] Sapsford RR, Hodges PW. The effect of abdominal and pelvic floor muscle activation on urine flow in women. Int Urogynecol J. 2012 Sep;23(9):1225-30. doi: 10.1007/s00192-011-1654-2. Epub 2012 Jan 26. PMID 22278713
- [Background] Sapsford RR, Hodges PW. Contraction of the pelvic floor muscles during abdominal maneuvers. Arch Phys Med Rehabil. 2001 Aug;82(8):1081-8. doi: 10.1053/apmr.2001.24297. PMID 11494188
- [Background] Skoura A, Billis E, Andriopoulou M, Drakonaki E, Papanikolaou DT, Tsekoura M, Kortianou E, Maroulis I. Intra- and inter-tester reliability of diaphragm thickness and excursion measurements of healthy women using rehabilitative ultrasound imaging across novice examiners. Eur J Transl Myol. 2025 Dec 19;35(4):13907. doi: 10.4081/ejtm.2025.13907. Epub 2025 Oct 27. PMID 41147924
- [Background] Dimitriadis Z, Kapreli E, Strimpakos N, Oldham J. Respiratory weakness in patients with chronic neck pain. Man Ther. 2013 Jun;18(3):248-53. doi: 10.1016/j.math.2012.10.014. Epub 2012 Nov 28. PMID 23199797
- [Background] Janssens L, McConnell AK, Pijnenburg M, Claeys K, Goossens N, Lysens R, Troosters T, Brumagne S. Inspiratory muscle training affects proprioceptive use and low back pain. Med Sci Sports Exerc. 2015 Jan;47(1):12-9. doi: 10.1249/MSS.0000000000000385. PMID 24870567
- [Background] O'Sullivan PB, Beales DJ. Changes in pelvic floor and diaphragm kinematics and respiratory patterns in subjects with sacroiliac joint pain following a motor learning intervention: a case series. Man Ther. 2007 Aug;12(3):209-18. doi: 10.1016/j.math.2006.06.006. Epub 2006 Aug 17. PMID 16919496
- [Background] Calvo-Lobo C, Almazan-Polo J, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P, Rodriguez-Sanz D, Lopez-Lopez D. Ultrasonography comparison of diaphragm thickness and excursion between athletes with and without lumbopelvic pain. Phys Ther Sport. 2019 May;37:128-137. doi: 10.1016/j.ptsp.2019.03.015. Epub 2019 Mar 28. PMID 30954705
- [Background] Ziaeifar M, Sarrafzadeh J, Noorizadeh Dehkordi S, Arab AM, Haghighatkhah H, Zendehdel Jadehkenari A. Diaphragm thickness, thickness change, and excursion in subjects with and without nonspecific low back pain using B-mode and M-mode ultrasonography. Physiother Theory Pract. 2022 Nov;38(13):2441-2451. doi: 10.1080/09593985.2021.1926022. Epub 2021 Jun 1. PMID 34061721
- [Background] Mohan V, Paungmali A, Sitilerpisan P, Hashim UF, Mazlan MB, Nasuha TN. Respiratory characteristics of individuals with non-specific low back pain: A cross-sectional study. Nurs Health Sci. 2018 Jun;20(2):224-230. doi: 10.1111/nhs.12406. Epub 2018 Feb 8. PMID 29421851
- [Background] Kharaji G, ShahAli S, Ebrahimi Takamjani I, Kashanian M, Sarrafzadeh J, Shanbehzadeh S. Ultrasound assessment of the abdominal, diaphragm, and pelvic floor muscles during the respiratory and postural tasks in women with and without postpartum lumbopelvic pain: a case-control study. Int Urogynecol J. 2023 Dec;34(12):2909-2917. doi: 10.1007/s00192-023-05621-2. Epub 2023 Aug 10. PMID 37561174
- [Background] Denizoglu Kulli H, Gurses HN. Relationship between inter-recti distance, abdominal muscle endurance, pelvic floor functions, respiratory muscle strength, and postural control in women with diastasis recti abdominis. Eur J Obstet Gynecol Reprod Biol. 2022 Dec;279:40-44. doi: 10.1016/j.ejogrb.2022.10.001. Epub 2022 Oct 5. PMID 36242869
- [Background] Koo P, Gartman EJ, Sethi JM, McCool FD. Physiology in Medicine: physiological basis of diaphragmatic dysfunction with abdominal hernias-implications for therapy. J Appl Physiol (1985). 2015 Jan 15;118(2):142-7. doi: 10.1152/japplphysiol.00276.2014. Epub 2014 Nov 6. PMID 25377882
- [Background] Marugan-Rubio D, Chicharro JL, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Rodriguez-Sanz D, Vicente-Campos D, Molina-Hernandez N, Calvo-Lobo C. Effectiveness of Ultrasonography Visual Biofeedback of the Diaphragm in Conjunction with Inspiratory Muscle Training on Muscle Thickness, Respiratory Pressures, Pain, Disability, Quality of Life and Pulmonary Function in Athletes with Non-Specific Low Back Pain: A Randomized Clinical Trial. J Clin Med. 2022 Jul 25;11(15):4318. doi: 10.3390/jcm11154318. PMID 35893409